CLINICAL TRIAL: NCT05324150
Title: M Charts Versus Amsler Test in Evaluating Metamorphopsia in Neovascular AMD Patients Treated With Anti-VEGF
Brief Title: M Charts Versus Amsler Test in Evaluating Metamorphopsia in nAMD
Acronym: MVAinAMD2022
Status: Completed | Type: Observational
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Andrea Greco, MD, Principal Investigator, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: Metamorphopsia_01
Record Dates: First submitted 2022-03-27; First posted 2022-04-12 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Macular Degeneration, Wet; Metamorphopsia
Keywords: Macular Degeneration Wet; nAMD; Metamorphopsia; Anti-VEGF Intravitreal Injections; Amsler Test; M Charts
MeSH Terms: conditions — Wet Macular Degeneration; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Age-related macular degeneration (AMD) is a complex eye disorder and the most common macular disease affecting millions of aged people in the developed countries, with an estimation that the number of AMD patients will be increased to 196 million in 2020, 288 million in 2040. Vision loss, central scotomas and metamorphopsia are the hallmark signs in patients with macular diseases. Metamorphopsia can be defined as a deformation of seen rectilinear lines due to photoreceptor separation/location and it is a typical but not exclusive sign of retinal disease. The most effective method of treating wet AMD is currently the anti-vascular endothelial growth factor intravitreal injections (anti-VEGF).

A further concern is the enormous costs and restriction of human resources that make periodic imaging unfeasible. Therefore, in patients with AMD treated by intravitreal anti-VEGF, monitoring with sensitive psychophysical tools could advance the time for diagnosis of CNV reactivation and enhance the outcome of treatment.

For assessment of the visual function, visual acuity and Amsler grid have been the gold standard. The Amsler grid is a simple and noninvasive test effortlessly understood by the patient, consisting of evenly spaced vertical and horizontal lines outlining 400 square, it has been widely adopted as a subjective test for metamorphopsia. However, it also produces high false-negative rate. Moreover, the answer to this test is dichotomous: straight or crooked lines and does not allow for quantification thus, it is problematic to monitor the visual function along the course and to evaluate the effectiveness of treatment with anti-VEGF agents. The M-chart (Inami Co., Tokyo, Japan) is a diagnostic device developed by Matsumoto to quantify the grade of metamorphopsia in patients with various types of macular diseases.

The usefulness of M-charts has been already demonstrated in different retinal diseases from macular pucker to BRVO.

The aim of this study is to compare the traditional Amsler grid and the M-Charts in evaluating metamorphopsia in patients suffering from wet AMD before and after Anti VEGF injection; and to match it with OCT results.

DETAILED DESCRIPTION:
Introduction

Age-related macular degeneration (AMD) is a complex eye disorder and the most common macular disease affecting millions of aged people in developed countries, with an estimation that the number of AMD patients will be increased to 196 million in 2020, 288 million in 2040. Vision loss, central scotomas, and metamorphopsia are the hallmark signs in patients with macular diseases. Metamorphopsia can be defined as a deformation of seen rectilinear lines due to photoreceptor separation/location and it is a typical but not exclusive sign of retinal disease. The most effective method of treating wet AMD is currently the anti-vascular endothelial growth factor intravitreal injections (anti-VEGF). Fluorescein angiography (FA) could be crucial for diagnosis but may be associated with serious complications, hence it has been replaced in clinical practice by Optical Coherence Tomography (OCT).

OCT is a quick and non-invasive procedure proving to be a detailed and reproducible tool for qualitative and quantitative assessment of the macular structure, and a useful tool for investigating the efficacy of anti-VEGF treatments in AMD patients. A further concern is the enormous costs and restriction of human resources that make periodic FA and OCT imaging unfeasible. Therefore, in patients with AMD treated by intravitreal anti-VEGF, monitoring with sensitive psychophysical tools could advance the time for diagnosis of CNV reactivation and enhance the outcome of treatment. For assessment of the visual function, visual acuity and Amsler grid have been the gold standard. The Amsler grid is a set of 7 charts of which the number one is the most commonly used: it a simple and noninvasive test effortlessly understood by the patient, consisting of evenly spaced vertical and horizontal lines outlining 400 square, it has been widely adopted as a subjective test for metamorphopsia. However, it also produces a decent false-negative rate. Moreover, the answer to this test is dichotomous: straight or crooked lines and does not allow for quantification thus, it is problematic to monitor the visual function along the course and to evaluate the effectiveness of treatment with anti-VEGF agents. The M-chart (Inami Co., Tokyo, Japan) is a diagnostic device developed by Matsumoto to quantify the grade of metamorphopsia in patients with various types of macular diseases.

The usefulness of M-charts has been already demonstrated in different retinal diseases from macular pucker to BRVO.

The aim of this study is to compare the traditional Amsler grid and the M-Charts in evaluating metamorphopsia in patients suffering from wet AMD before and after Anti VEGF injection, and to match it with OCT results.

Methods An expected total of 150 patients will be selected prospectively from the retinal out-patient clinic of the Ophthalmology Department in Cuneo, Italy. The study is approved by the independent ethics committee and performed in accordance with the Declaration of Helsinki. A written informed consent will be required from each participant after the explanation of the nature of the study together with the intravitreal one. Patients at their first wet AMD diagnosis by means of FA and with a best-corrected visual acuity, better than or equal to 1.0 logMAR will be involved in the study and included in a loading phase with three IVT injections spaced one month one from the other in a treat and extend protocol fashion. Inclusion criteria will be a diagnosis of neovascular age-related macular degeneration with active CNV on fluorangiographic examination, visual acuity equal or greater than 1.0 logMAR written informed consent, age over 50.

The exclusion criteria will be prior intravitreal injection, intraocular surgery, major ocular diseases such as amblyopia, glaucoma, or strabismus, and refracting errors greater than 4D. The first and the follow-up examination performed at one, three, six and twelve months later will include a comprehensive ophthalmological examination (slit-lamp examination, applanation tonometry, dilated funduscopy) and OCT (Heidelberg Engineering,Germany). Visual acuity will be tested using ETDRS and the Amsler chart ( Chart 1 black grid on white background) with undilated pupils and the best near correction. The M-charts consist of 19 dotted lines subtending 20° at 30 cm in which the dot separation varies systematically from 0.2° to 2°: with coarser sampling, the perception of metamorphopsia is reduced and in some cases negated. The examiner will present consecutive dotted lines, starting with a solid line (0) and the patient has to state whether the conferred line is distorted or not. When the patient recognizes the dotted line presented as being straight, its visual angle is counted to be the metamorphopsia score. M-charts are rotated by 90 degrees for both vertical (VM) and horizontal presentation (HM). Central retinal thickness (CRT) will be collected as a quantitative parameter, and for the morphological part, the nAMD will be subdivided in CNV type I or II with additional information on the presence of sub-retinal fluid (SRF), intraretinal-fluid (IRF), and epithelial detachment. For the present study, only one eye of each patient will be taken into consideration. The injections are gonna be performed in an operating room via pars plana following the most recent expert consensus recommendations on IVI techniques.

Statistical analysis The Amsler test will be considered positive whenever a distorted view of the lines. The M-charts test will be considered positive if the metamorphopsia has a score greater than 0, where 0 is considered a negative result. This evaluation will be done separately in relation to the horizontal (HM) and vertical (VM) parameters. Not assuming a normal distribution sample, the Kruskal Wallis test will be used to compare the median values of VM and HM and visual acuity expressed in LogMAR and the thickness value central retinal (CRT) before and after intravitreal injections of Anti-VEGF in the three groups.Spearman's correlation coefficient will be used to evaluate the relationship between metamorphopsia, visual acuity and the CRT. The Anova mixed-model test will be used to determine the effect of time in different measurements. The level of statistical significance reported is P 0.05, while sensitivity and specificity will be calculated with the 95% confidence interval.The data for statistical analysis will be collected with (Microsoft Excel 2007; Microsoft Inc., Redmond,WA), and calculated with Statistical Package for Social Sciences (version 17.0, SPSS Inc., Chicago, IL).

Conclusion The goal of this study will be to compare the results of the classic Amsler grid and the less known M-charts with OCT results in the evaluation of metamorphopsia in wet AMD patient treated with the three main one's IVT drugs. The best current practice involves using the Amsler charts for detecting and monitoring metamorphopsia in AMD, but more than one study has shown limitations regarding this exam, including false positives, dichotomous response and false negatives.

There are many possible explanations for the false-negative rate: firstly, the filling-in phenomenon across pathological scotomas; secondly, the use of a preferred retinal locus away from the scotoma boundary moreover, probably, the averaging of crowded stimuli, the results of the Amsler charts are only descriptive; they are neither precise nor reproducible. Thus the Amsler chart alone does not seem to be sufficient for the metamorphopsia detection and for monitoring the changes over time.It has been demonstrated that the M-charts may be used as a diagnostic tool in the detection of metamorphopsia in AMD patients. The rate of metamorphopsia detection in patients addressed to the intravitreal injection was higher with the M-charts (89%) than with Amsler test (69%) in a study. Thus, it seems that the M-charts are superior to the Amsler grid in detecting metamorphopsia in patients with wet AMD. In the current study, the investigator want to show that with the M-charts, it is possible to monitor quantitatively the changes in the degree of metamorphopsia over time.

As far as the investigators know this research will be the first to compare the degree of metamorphopsia between 3 different drugs used in nAMD, and for an intermediate period of twelve months.

Other authors have reported the modification of metamorphopsia after one month of follow up and with bevacizumab alone.

The M-charts provide repeatable clinical information regarding metamorphopsia, another feature of the visual function, that seems independent from visual acuity and OCT results. Plus it could become an additional parameter for the prognostic evaluation of clinical efficacy of intravitreal injections in patients with nAMD. Patient Satisfaction under IVT treatment for wet AMD may be not necessarily measured by BCVA alone. Therefore, evaluating both the MH and MV scores in addition to BCVA can be an independent treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration with active CNV on fluorangiographic examination
* Visual acuity (VA) equal to or greater than 1.0 logMAR
* Written informed consent
* Age over 50.

Exclusion Criteria:

* Prior intravitreal injection or intraocular surgery
* Major ocular diseases such as amblyopia, glaucoma, or strabismus, and refracting errors greater than 4D.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Case only study: heterogeneous group of patients diagnosed with active maculopathy
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in VM | baseline and after 1, 3, 6, 12 months ( 5 measurements)
  Change in values of Vertical M Charts ( from 0 to 2.0 )
Change in HM | baseline and after 1, 3, 6, 12 months ( 5 measurements)
  Change in values of Horizontal M Charts ( from 0 to 2.0)
Change in Amsler Test | baseline and after 1, 3, 6, 12 months ( 5 measurements)
  Change in values of this test: Positivity (+) or negativity (-)

SECONDARY OUTCOMES:
CRT | baseline, after 1, 3, 6, 12 months
  Central Retinal Thickness at OCT scan
Visual Acuity | baseline, after 1, 3, 6, 12 months
  Visual Acuity on LogMAR scale

OTHER OUTCOMES:
OCT morphological parameters | baseline, after 1, 3, 6, 12 months
  Presence of SRF, IRF and epitelial Detachment in CNV ( type I or II)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Violante, MD, Study Chair — OSCroceCarle, +39 0171 641571
Locations (1):
- Ospedale Santa Croce, Cuneo, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Simunovic MP. METAMORPHOPSIA AND ITS QUANTIFICATION. Retina. 2015 Jul;35(7):1285-91. doi: 10.1097/IAE.0000000000000581. PMID 26049620
- [Background] Campa C, Parodi MB. Anti-Vegf Therapy for Ocular Diseases: Present and Future. Curr Drug Targets. 2020;21(12):1158. doi: 10.2174/138945012112200727153907. No abstract available. PMID 32957867
- [Background] Musa F, Muen WJ, Hancock R, Clark D. Adverse effects of fluorescein angiography in hypertensive and elderly patients. Acta Ophthalmol Scand. 2006 Dec;84(6):740-2. doi: 10.1111/j.1600-0420.2006.00728.x. PMID 17083530
- [Background] Loewenstein A, Malach R, Goldstein M, Leibovitch I, Barak A, Baruch E, Alster Y, Rafaeli O, Avni I, Yassur Y. Replacing the Amsler grid: a new method for monitoring patients with age-related macular degeneration. Ophthalmology. 2003 May;110(5):966-70. doi: 10.1016/S0161-6420(03)00074-5. PMID 12750099
- [Background] Wada I, Yoshida S, Kobayashi Y, Zhou Y, Ishikawa K, Nakao S, Hisatomi T, Ikeda Y, Ishibashi T, Sonoda KH. Quantifying metamorphopsia with M-CHARTS in patients with idiopathic macular hole. Clin Ophthalmol. 2017 Sep 20;11:1719-1726. doi: 10.2147/OPTH.S144981. eCollection 2017. PMID 29033537
- [Background] Nowomiejska K, Oleszczuk A, Brzozowska A, Grzybowski A, Ksiazek K, Maciejewski R, Ksiazek P, Juenemann A, Rejdak R. M-charts as a tool for quantifying metamorphopsia in age-related macular degeneration treated with the bevacizumab injections. BMC Ophthalmol. 2013 Apr 15;13:13. doi: 10.1186/1471-2415-13-13. PMID 23587218
- [Background] Querques G, Querques L, Rafaeli O, Canoui-Poitrine F, Bandello F, Souied EH. Preferential hyperacuity perimeter as a functional tool for monitoring exudative age-related macular degeneration in patients treated by intravitreal ranibizumab. Invest Ophthalmol Vis Sci. 2011 Sep 1;52(9):7012-8. doi: 10.1167/iovs.11-7517. PMID 21885622
- [Background] Schuchard RA. Validity and interpretation of Amsler grid reports. Arch Ophthalmol. 1993 Jun;111(6):776-80. doi: 10.1001/archopht.1993.01090060064024. PMID 8512478